CLINICAL TRIAL: NCT04422119
Title: Standard Dressing Versus Moist Dressing in the Course of the Postoperative Wound in Patients With Knee Prosthesis
Acronym: APOSIT-PTG
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Germans Trias i Pujol Hospital (Other)
Collaborators: Fundació Institut Germans Trias i Pujol (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: AC-16-016-CEIMPS
Record Dates: First submitted 2019-12-03; First posted 2020-06-09 (Actual); Last update posted 2020-06-09 (Actual); Status verified 2020-06

CONDITIONS: Surgical Wound; Knee Disease
Keywords: Surgical wound healing; knee arthroplasty; postoperative dressings
MeSH Terms: conditions — Surgical Wound

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Multi-layer foam dressing (Experimental): Patients in experimental group will receive the application of a multi-layer foam dressing with Safetac in surgical wound
  Interventions: Procedure: Multi-Foam dressing
- Usual care (Active Comparator): Patients in control group will receive standard treatment with povidone-iodine and a gauze dressing with plaster.
  Interventions: Procedure: Usual care

INTERVENTIONS:
Procedure: Multi-Foam dressing — Application of a multi-layer foam dressing with Safetac in surgical wound
  Arms: Multi-layer foam dressing
Procedure: Usual care — Care of surgical wound with povidone-iodine and a gauze dressing with plaster.
  Arms: Usual care

SUMMARY:
The aim of the study is: to evaluate the efficacy of two post-operative dressings in the management of the surgical wounds in patients who received a knee prosthesis

DETAILED DESCRIPTION:
This was a randomised, controlled, clinical trial on patients who received a primary knee prosthesis in 2018-2019. Treatment group was given a multi-layer foam dressing with Safetac. The control group received standard treatment with povidone-iodine and a gauze dressing with plaster. 50 patients was needed for sufficient power. Primary outcome measures were; the characteristics of the surgical wound, patient reported comfort and adaptability according to the physiotherapist. Secondary outcome measures were: the clinical status and quality of life level according to the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC). Statistical analysis was performed by using IBM SPSS version 25, with a statistical significance of 5%.

ELIGIBILITY:
Inclusion Criteria:

* Surgical intervention of total primary knee prosthesis
* Informed consent approved and signed by participants.

Exclusion Criteria:

* Sensitivity or allergy to study dressings

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2018-06-01 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Change in number of dressing changes | From fist day post-surgery to 7th postoperative day
  Number of dressing applications to the patients required

SECONDARY OUTCOMES:
Change in patient comfort | From fist day post-surgery to 7th postoperative day
  Patient comfort reported in a scale from 1 (non satisfactory) - to 4 (very satisfactory)

CONTACTS AND LOCATIONS:
Overall Officials: Antonia Salmerón-Ramírez, RN, Principal Investigator — Germans Trias i Pujol Hospital
Locations (1):
- Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No